CLINICAL TRIAL: NCT06797895
Title: Designing a Virtual Reality Intervention to Improve Physical and Psychological Health in Intensive Care Units
Acronym: GAMERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00116448
Record Dates: First submitted 2024-12-09; First posted 2025-01-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-01

CONDITIONS: Mobility; ICU; Heart Surgery; Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality (VR) intervention (Other): Cohort for observing the effects of the VR intervention on ICU mobility.
  Interventions: Behavioral: VR assisted mobility

INTERVENTIONS:
Behavioral: VR assisted mobility — Commercially-based VR experience used to help move upper extremities to music, similar to dancing or Tai-Chi.

SUMMARY:
The goal of this study is to explore if Virtual Reality helps patients in the cardiothoracic ICU move more and feel better. Participants will be asked to answer a survey about anxiety, depression, and loneliness. The study team will teach participants how to use the VR device and how to play the game. Participants will play the game at least once per day, but can play as much as they want. Study activities include nurse facilitated patient use of VR applications that involve upper body movement (e.g., using arms and hands to dance or hit objects in a virtual reality environment).

DETAILED DESCRIPTION:
Patients who survive critical illness and prolonged intensive care unit (ICU) stays are at risk for debilitating physical (deconditioning, skin injury, and infection), and mental health impairment (depression, anxiety and PTSD). Early mobility improves these deleterious outcomes but is challenging to implement in patients on prolonged bedrest. The purpose of this study is to compare a nurse-led implementation of a Virtual Reality (VR) experience in the Cardio-Thoracic Intensive Care Unit (CT-ICU) to standard of care to improve mobility for patients on prolonged bedrest. The investigators hypothesize that nurse-led implementation of VR experiences in the CT-ICU, in combination with engineering-led patient-centered customization of the VR applications, will improve both the physical and psychological function of ICU patients on prolonged bedrest.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* English speaking
* 3+ days ICU admission with limited mobility

Exclusion Criteria:

* Pregnancy
* Blind/severe visual impairment
* History of seizures
* Intubation/sedation
* Special enteric contact isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by nursing time required | up to 6 months
  For each participant, the total nursing time spent (in minutes) setting up and delivering the intervention will be recorded.

SECONDARY OUTCOMES:
Usability as measured by patient-reported ease of playing the game | up to 6 months
  Usability: Using a 5-point Likert scale (0- very difficult to 5- very easy; higher is better outcome), participants will be surveyed after the intervention period to assess ease of playing the game.
Usability as measured by patient-reported ease of hand controller use | up to 6 months
  Usability: Using a 5-point Likert scale (0- very difficult to 5- very easy; higher is better outcome), participants will be surveyed after the intervention period to assess ease of hand controller use.
Usability as measured by patient-reported wearability of headset | up to 6 months
  Usability: Using a 5-point Likert scale (0- very difficult to 5- very easy; higher is better outcome), participants will be surveyed after the intervention period to assess wearability of headset.
Usability as measured by patient-reported comfort of headset | up to 6 months
  Usability: Using a 5-point Likert scale (0- very difficult to 5- very easy; higher is better outcome), participants will be surveyed after the intervention period to assess comfort of headset.
Number of participants who find the intervention acceptable | up to 6 months
  Acceptability: Participants will be asked if they would recommend this game to a friend or loved one, yes or no.
Change in mobility activity frequency | Baseline, 6 months
  To determine if a VR intervention increases mobility for patients on prolonged bedrest, the frequency of VR sessions is recorded. Frequency will be reported as counts.
Change in mobility activity time | Baseline, 6 months
  To determine if a VR intervention increases mobility for patients on prolonged bedrest, the duration of each VR session is recorded. Activity will be reported as total minutes.
Change in Hospital Anxiety and Depression Scale (HADS) - anxiety | Baseline to day 10 or ICU transfer, whichever comes first
  The Hospital Anxiety and Depression Scale (HADS) is a self-report scale used to measure the severity of depression and anxiety in patients with comorbid medical conditions. The total score for anxiety ranges from 0 to 21, where a higher score indicates greater anxiety.
Change in Hospital Anxiety and Depression Scale (HADS) - depression | Baseline to day 10 or ICU transfer, whichever comes first
  The Hospital Anxiety and Depression Scale (HADS) is a self-report scale used to measure the severity of depression and anxiety in patients with comorbid medical conditions. The total score for depression ranges from 0 to 21, where a lower score indicates greater depression.
Change in UCLA 3-item Loneliness Scale | Baseline to day 10 or ICU transfer, whichever comes first
  This scale comprises 3 questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation. The total score ranges from 0 to 9, where a higher score indicates greater loneliness.

OTHER OUTCOMES:
Change in BDNF (brain-derived neurotrophic factor) level | Baseline to day 10 or ICU transfer, whichever comes first
  BDNF may play a role in the biology of mood disorders.
Change in TNF (tumor necrosis factor) level | Baseline to day 10 or ICU transfer, whichever comes first
  TNF is a protein that plays a role in the development of depression and other psychiatric disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Mall, MSN, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No